CLINICAL TRIAL: NCT02762019
Title: LAMPO: Multicenter Randomized Double-blind Controlled Trial to Evaluate the Efficacy of Laser Therapy for Treatment of Oral Mucositis Induced by Chemotherapy in Children
Brief Title: Laser for Oral Mucositis in Pediatric Onco-hematology
Acronym: LAMPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC 33/12
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Stomatitis
Keywords: Stomatitis; Laser; Children; Chemotherapy; Treatment
MeSH Terms: conditions — Stomatitis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser therapy (Experimental): Children are allocated to receive Laser therapy
  Interventions: Device: Laser therapy
- Sham therapy (Sham Comparator): Children are allocated to receive Sham therapy
  Interventions: Device: Sham therapy

INTERVENTIONS:
Device: Laser therapy — Treatment with K-Laser Cube3 during 4 consecutive days, with the following protocol: 660-970 nm wavelength, 3,2W mean power (6.4W pulsating at 50%), 3'51'' duration, 1-20000 Hz frequency, and 1 cm2 spot size. Laser application was performed all over the oral cavity.
  Arms: Laser therapy
Device: Sham therapy — Only the laser pointer movement, without laser activation, during 4 consecutive days, all over the oral cavity.
  Arms: Sham therapy

SUMMARY:
Children with cancer undergoing intensive chemotherapy (CT) regimens experience many side effects among which oral mucositis (OM) is one of the most debilitating. Modifications of CT's schedule and prolonged hospitalization may be necessary in presence of OM, causing poor general conditions and debilitation. Moreover, the use of narcotic analgesics and total parenteral nutrition may be required, triggering not only a physical deficit but also an economic burden. Despite the frequency and impact of OM among children with cancer, there is no consensus on standard therapy for this condition. Previous studies demonstrated that high power laser therapy can help the maintenance of nutritional status in patients with OM and can remarkably reduce costs/resources needed. Laser therapy has evidence of efficacy in reducing symptoms and in preventing the onset of OM in adult cancer patients but only one randomized controlled trial, with a limited number of children enrolled, supports its use in children for treatment of OM induced by chemotherapy.

This multicenter double-blind randomized controlled trial evaluates the efficacy of laser for treatment of oral mucositis secondary to chemotherapy in children aged 3-17 years.

The study involves 8 italian hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-18 years
* Oral mucositis of grade 3 or 4 at enrollment (CTC - WHO scale)
* Antiblastic chemotherapy in the in the previous three weeks
* Willingness to undergo treatment for 4 consecutive days and to return for evaluation 7 and 11 days after enrollment.

Exclusion Criteria:

* Previous treatment with laser therapy for stomatitis
* Presence of dysplastic oral lesions
* Reduction of mouth opening (<1 cm)
* Localized head and/or neck radiation treatment in the previous 4 weeks
* Use of keratinocyte growth factor (KGF)
* Previous enrollment in the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the grade of oral mucositis | 7 days after enrollment
  Reduction of stomatitis' grade (from grade 3 or 4 to a lower grade). The grade of stomatitis is defined using the World Health Organization (WHO) evaluation scale

SECONDARY OUTCOMES:
Reduction of the grade of oral mucositis | 3 days after enrollment
  Reduction of stomatitis' grade (from grade 3 or 4 to a lower grade). The grade of stomatitis is defined using the WHO evaluation scale
Reduction of the grade of oral mucositis | 11 days after enrollment
  Reduction of stomatitis' grade (from grade 3 or 4 to a lower grade). The grade of stomatitis is defined using the WHO evaluation scale
Reduction of pain, age 4-7 years | 3 days after enrollment
  Reduction of self-reported pain recorded with the Faces Pain Scale-Revised (FPS-R)
Reduction of pain, age 8-18 years | 3 days after enrollment
  Reduction of self-reported pain recorded with a numeric rating scale
Reduction of pain, age 4-7 years | 7 days after enrollment
  Reduction of self-reported pain recorded with the Faces Pain Scale-Revised (FPS-R)
Reduction of pain, age 8-18 years | 7 days after enrollment
  Reduction of self-reported pain recorded with a numeric rating scale
Reduction of pain, age 4-7 years | 11 days after enrollment
  Reduction of self-reported pain recorded with the Faces Pain Scale-Revised (FPS-R)
Reduction of pain, age 8-18 years | 11 days after enrollment
  Reduction of self-reported pain recorded with a numeric rating scale
Reduction of need for analgesics | at day 7
Adverse events | at day 11

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Andrea Zanazzo, MD, Study Chair — IRCCS Burlo Garofolo, Trieste; Matteo Biasotto, DDS, Study Chair — Azienda Ospedaliero Universitaria "Ospedali Riuniti", Trieste
Locations (8):
- Italy (8):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Spedali civili Ospedale dei Bambini, Brescia
  - Ospedale Pediatrico Microcitemico "Antonio Cao", Cagliari
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero universitaria di Parma, Parma
  - Fondazione IRCCS, Policlinico San Matteo, Pavia
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - IRCCS Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: Undecided